CLINICAL TRIAL: NCT03669211
Title: A Pilot, Prospective Study Assessing the Evolution of Cardiovascular Function and Quality of Life in Patients With Acute Coronary Syndrome, Included in the SCArabée Therapeutic Education Program
Brief Title: Evolution of Cardiovascular Function and Quality of Life in Patients Included in the SCArabée Therapeutic Education Program
Acronym: SCArabée
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Mutualiste de Grenoble (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018/06-JPE-GHMG
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Acute Coronary Syndrome
Keywords: Therapeutic education; Cardiac stress test
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac stress test (Experimental)
  Interventions: Diagnostic Test: Cardiac stress test

INTERVENTIONS:
Diagnostic Test: Cardiac stress test — In order to assess the evolution of their cardiorespiratory function, patients will benefit from two cardiac stress test combined with VO2 study, one at inclusion in the study, and the other one 6 months later.
  Other Names: Cardiac diagnostic test; Cardiopulmonary exercise test; CPX test

SUMMARY:
Coronary artery disease is defined as a disease of the arteries that vascularize the heart, resulting in myocardial ischemia, i.e. insufficient blood supply to the heart muscle. Eventually, it may be responsible for acute coronary syndrome that includes unstable angina (chest pain) and myocardial infarction (necrosis of the heart muscle).

The main cause of this disease is atheroma, and management involves reducing modifiable cardiovascular risk factors (sedentary lifestyle, smoking, obesity, high blood pressure, diabetes, dyslipidemia). Every year, this disease affects more than 120 000 people in France, aging 65 years on average.

In this real public health problem, there is a significant discrepancy between the excellence of the management of the acute incident and the inadequacy of the re-adaptive and educational management of the care suites. In fact, it is noted that hospitalization times are short given the progress of myocardial revascularization, associated with a low intra-hospital mortality rate, 3% but the places in rehabilitation programs ("Soins de Suite et de Réadaptation" or "SSR") are too limited (25% of the patients are included in these programs). Physical rehabilitation has proven effective for decades, with robust evidence of decreased recurrence and mortality (-20%).

At the Groupe Hospitalier Mutualiste of Grenoble, France, patients are offered two courses of treatment in post-myocardial infarction:

* A therapeutic education program: SCarabée,
* A rehabilitation program (SSR) The therapeutic education program aims to help the patient identify his needs, acquire knowledge, strengthen his resources and finally develop with him a project to improve his quality of life.

SSR offers physical rehabilitation as a treatment for infarction, which improves cardiovascular function, which is assessed by the cardiorespiratory test.

Is the Scarabée therapeutic education program is sufficient to help the patient improve his physical abilities? This study aims to answer this question, by setting up a reinforced monitoring of the evolution of the cardiovascular function of the patients included in the SCArabée program, via cardiorespiratory tests. The results of this first pilot study will potentially lead to a second randomized study comparing therapeutic education associated with Adapted Physical Education versus therapeutic education alone for the improvement of cardiorespiratory functions and the quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 or older
* Patient with newly diagnosed or recurring Acute Coronary Syndrome, or presenting a coronary heart disease detected on ischemia test and stented
* Patient included in the SCArabée therapeutic education program
* Patient assessed stable on the basis of a clinical examination, or exercise test, or ultrasound data
* Patient in physical capacity to perform a cardiorespiratory test
* Patient giving free, informed and written consent
* Patient affiliated to the social security system

Exclusion Criteria:

* Impossibility to submit to follow-up of the study for geographical social or psychological reasons
* Persons referred to in Articles L1121-5 to L1121-8 of the Public Health Code (corresponds to all persons protected): pregnant woman, parturient, nursing mother, person deprived of liberty by judicial or administrative decision, person making the subject of a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Assess the evolution of cardiovascular function of patients included in the SCArabée program | At inclusion, and 6 month after inclusion
  Endpoint : Percentage change in the VO² threshold between the two cardiac stress tests

SECONDARY OUTCOMES:
Assess the evolution of the patient's physical activity | At inclusion, and 6 month after inclusion
  Endpoint : Score of the "Ricci and Gagnon" questionnaire filled by the patient
Assess the evolution of cardiac function | At inclusion, and 6 month after inclusion
  Endpoint : Left Ventricular Ejection Fraction measured during the two cardiac stress tests
Assess the evolution of perceived level of anxiety | At inclusion, and 6 month after inclusion
  Endpoint : Score of the Hospital Anxiety and Depression Scale filled by the patient
Assess the evolution of global quality of life | At inclusion, and 6 month after inclusion
  Endpoint : Score of the 12-Item Short Form Health Survey (SF-12) filled by the patient
Assess the evolution of weight | At inclusion, and 6 month after inclusion
  Measured during a bioelectrical impedance analysis
Assess the evolution of fat mass | At inclusion, and 6 month after inclusion
  Measured during a bioelectrical impedance analysis
Assess the evolution of visceral fat mass | At inclusion, and 6 month after inclusion
  Measured during a bioelectrical impedance analysis
Assess the evolution of muscular mass | At inclusion, and 6 month after inclusion
  Measured during a bioelectrical impedance analysis
Assess the evolution of Body Mass Index | At inclusion, and 6 month after inclusion
Assess the evolution of tobacco consumption | At inclusion, and 6 month after inclusion
  Comparison of the number of cigarettes consumed per day between the month preceeding the Acute Coronary Syndrome event and the 6th month of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Mutualiste de Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Puymirat E, Simon T, Cayla G, Cottin Y, Elbaz M, Coste P, Lemesle G, Motreff P, Popovic B, Khalife K, Labeque JN, Perret T, Le Ray C, Orion L, Jouve B, Blanchard D, Peycher P, Silvain J, Steg PG, Goldstein P, Gueret P, Belle L, Aissaoui N, Ferrieres J, Schiele F, Danchin N; USIK, USIC 2000, and FAST-MI investigators. Acute Myocardial Infarction: Changes in Patient Characteristics, Management, and 6-Month Outcomes Over a Period of 20 Years in the FAST-MI Program (French Registry of Acute ST-Elevation or Non-ST-Elevation Myocardial Infarction) 1995 to 2015. Circulation. 2017 Nov 14;136(20):1908-1919. doi: 10.1161/CIRCULATIONAHA.117.030798. Epub 2017 Aug 27. PMID 28844989
- [Background] Kotseva K, De Bacquer D, De Backer G, Ryden L, Jennings C, Gyberg V, Abreu A, Aguiar C, Conde AC, Davletov K, Dilic M, Dolzhenko M, Gaita D, Georgiev B, Gotcheva N, Lalic N, Laucevicius A, Lovic D, Mancas S, Milicic D, Oganov R, Pajak A, Pogosova N, Reiner Z, Vulic D, Wood D, On Behalf Of The Euroaspire Investigators. Lifestyle and risk factor management in people at high risk of cardiovascular disease. A report from the European Society of Cardiology European Action on Secondary and Primary Prevention by Intervention to Reduce Events (EUROASPIRE) IV cross-sectional survey in 14 European regions. Eur J Prev Cardiol. 2016 Dec;23(18):2007-2018. doi: 10.1177/2047487316667784. Epub 2016 Sep 27. PMID 27638542
- [Background] Belle L, Cayla G, Cottin Y, Coste P, Khalife K, Labeque JN, Farah B, Perret T, Goldstein P, Gueugniaud PY, Braun F, Gauthier J, Gilard M, Le Heuzey JY, Naccache N, Drouet E, Bataille V, Ferrieres J, Puymirat E, Schiele F, Simon T, Danchin N; FAST-MI 2015 investigators. French Registry on Acute ST-elevation and non-ST-elevation Myocardial Infarction 2015 (FAST-MI 2015). Design and baseline data. Arch Cardiovasc Dis. 2017 Jun-Jul;110(6-7):366-378. doi: 10.1016/j.acvd.2017.05.001. Epub 2017 Jun 21. PMID 28647465
- [Background] Fox KA, Carruthers KF, Dunbar DR, Graham C, Manning JR, De Raedt H, Buysschaert I, Lambrechts D, Van de Werf F. Underestimated and under-recognized: the late consequences of acute coronary syndrome (GRACE UK-Belgian Study). Eur Heart J. 2010 Nov;31(22):2755-64. doi: 10.1093/eurheartj/ehq326. Epub 2010 Aug 30. PMID 20805110
- [Background] Pavy B, Barbet R, Carre F, Champion C, Iliou MC, Jourdain P, Juilliere Y, Monpere C, Brion R; Working Group of Exercise Rehabilitation and Sport; Therapeutic Education Commission of the French Society of Cardiology. Therapeutic education in coronary heart disease: position paper from the Working Group of Exercise Rehabilitation and Sport (GERS) and the Therapeutic Education Commission of the French Society of Cardiology. Arch Cardiovasc Dis. 2013 Dec;106(12):680-9. doi: 10.1016/j.acvd.2013.10.002. Epub 2013 Nov 15. PMID 24239052
- [Background] Nocon M, Hiemann T, Muller-Riemenschneider F, Thalau F, Roll S, Willich SN. Association of physical activity with all-cause and cardiovascular mortality: a systematic review and meta-analysis. Eur J Cardiovasc Prev Rehabil. 2008 Jun;15(3):239-46. doi: 10.1097/HJR.0b013e3282f55e09. PMID 18525377
- [Background] Hambrecht R, Walther C, Mobius-Winkler S, Gielen S, Linke A, Conradi K, Erbs S, Kluge R, Kendziorra K, Sabri O, Sick P, Schuler G. Percutaneous coronary angioplasty compared with exercise training in patients with stable coronary artery disease: a randomized trial. Circulation. 2004 Mar 23;109(11):1371-8. doi: 10.1161/01.CIR.0000121360.31954.1F. Epub 2004 Mar 8. PMID 15007010
- [Background] Anderson L, Thompson DR, Oldridge N, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2016 Jan 5;2016(1):CD001800. doi: 10.1002/14651858.CD001800.pub3. PMID 26730878
- [Background] Wood DA, Kotseva K, Connolly S, Jennings C, Mead A, Jones J, Holden A, De Bacquer D, Collier T, De Backer G, Faergeman O; EUROACTION Study Group. Nurse-coordinated multidisciplinary, family-based cardiovascular disease prevention programme (EUROACTION) for patients with coronary heart disease and asymptomatic individuals at high risk of cardiovascular disease: a paired, cluster-randomised controlled trial. Lancet. 2008 Jun 14;371(9629):1999-2012. doi: 10.1016/S0140-6736(08)60868-5. PMID 18555911
- [Background] Giannuzzi P, Temporelli PL, Marchioli R, Maggioni AP, Balestroni G, Ceci V, Chieffo C, Gattone M, Griffo R, Schweiger C, Tavazzi L, Urbinati S, Valagussa F, Vanuzzo D; GOSPEL Investigators. Global secondary prevention strategies to limit event recurrence after myocardial infarction: results of the GOSPEL study, a multicenter, randomized controlled trial from the Italian Cardiac Rehabilitation Network. Arch Intern Med. 2008 Nov 10;168(20):2194-204. doi: 10.1001/archinte.168.20.2194. PMID 19001195
- [Background] Wasserman K, Hansen JE, Sue DY, Whipp BJ, Froelicher VF. Principles of Exercise Testing and Interpretation. Journal of Cardiopulmonary Rehabilitation and Prevention. avr 1987;7(4):189.
- [Background] Pavy B, Iliou MC, Meurin P, Tabet JY, Corone S; Functional Evaluation and Cardiac Rehabilitation Working Group of the French Society of Cardiology. Safety of exercise training for cardiac patients: results of the French registry of complications during cardiac rehabilitation. Arch Intern Med. 2006 Nov 27;166(21):2329-34. doi: 10.1001/archinte.166.21.2329. PMID 17130385
- [Background] Cerretelli P. Traité de physiologie de l'exercice et du sport. Elsevier Masson; 2002. 504 p.
- [Background] Wilmore JH, Costill DL, Kenney L. Physiologie du sport et de l'exercice. De Boeck Superieur; 2017. 644 p.